CLINICAL TRIAL: NCT00472186
Title: The Effects of Gastro-esophageal Acid Suppression on Post-tonsillectomy Pain
Brief Title: The Effects of Reducing Stomach Acid on Post-tonsillectomy Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor compliance with returning of logbooks by families. Two patients were enrolled. Only one returned the logbook and therefore not analyzed
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Manali Amin, Instructor, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 06-11-0513
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Results first posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Post-tonsillectomy Pain; Post-tonsillectomy Activity; Post-tonsillectomy Hydration
Keywords: Tonsillectomy; Pain
MeSH Terms: conditions — Pain | interventions — Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Post-operative administration of Lansoprazole
  Interventions: Drug: Lansoprazole
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lansoprazole — If weight is less than 30 kg, 15 mg of Lansoprazole twice daily will be administered. If weight is greater than or equal to 30 kg, 30 mg of Lansoprazole twice daily will be administered.
  Other Names: Prevacid
  Arms: 1
Drug: Placebo — Placebo will also be administered based on weight.
  Arms: 2

SUMMARY:
This study was designed to determine whether post-operative pain following a tonsillectomy can be reduced by adding an antacid-like medication to the medications taken after surgery. It is hypothesized that even a small amount of stomach acid backing up and entering the mouth can increase post-tonsillectomy pain. Therefore, the use of an antacid-like medication should help to decrease pain and reduce the amount of narcotic medication required for pain control.

DETAILED DESCRIPTION:
This study has been limited to children and adolescents ages 5-18 who are undergoing tonsillectomy for an indication of obstructive sleep disturbance (snoring, choking/gasping or pauses in breathing during sleep.)

Study participants will be randomized to two groups: study medication (Lansoprazole) or an inactive substance(placebo).

Participants will be asked to do all of the following:

1. Take the study medication twice a day for 14 days.
2. Keep a log book which will include:

   * Record the medications and amount of each medication taken each day for 14 days. This includes pain medication and the study drug.
   * Record your child's activity level daily for 14 days.
   * Collect your child's urine one time daily and test it using special medicated strips to monitor their daily liquid intake for 14 days.
3. Meet with a Research Assistant or Study Physician 14-21 days after the study to collect the log book and perform a post-operative examination.

ELIGIBILITY:
Inclusion Criteria:

* All healthy children ages 5-18 years scheduled for tonsillectomy and /or adenotonsillectomy for sleep disturbance secondary to airway obstruction at Children's Hospital Boston

Exclusion Criteria:

* Patients on any medications other than the study drug (Lansoprazole or placebo), Amoxicillin®, and acetaminophen with or without codeine
* An underlying medical condition which would necessitate an alteration in the anesthetic regimen
* Patients allergic to any of the medications in the protocol
* History of chronic tonsillitis
* History of chronic pain conditions
* History of active gastro-esophageal reflux disease
* Surgery in addition to tonsillectomy/adenotonsillectomy (except for myringotomy)
* Cognitive/developmental disorders
* Inability to use a self-report pain scale

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manali Amin, MD, Principal Investigator — Children's Hosptial Boston
Locations (2):
- United States (2):
  - Children's Hospital Boston, Boston, Massachusetts
  - Childrens Hospital Boston, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated due to low recruitment, since only one participant returned logbooks with data there are concerns with confidentiality therefore no data is being reported.
Groups:
- 1: Post-operative Administration of Lansoprazole: Lansoprazole: If weight is less than 30 kg, 15 mg of Lansoprazole twice daily will be administered. If weight is greater than or equal to 30 kg, 30 mg of Lansoprazole twice daily will be administered.
- 2: Placebo: Placebo: Placebo will also be administered based on weight.
Period: Overall Study
Arm/Group | 1: Post-operative Administration of Lansoprazole | 2: Placebo
Started | 2 | 0
Completed | 1 | 0
Not Completed | 1 | 0
Not completed — Study was terminated due to poor compliance with returning logbooks by families. | 1 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated due to low recruitment, since only one participant returned logbooks with data there are concerns with confidentiality therefore no data is being reported.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1: Post-operative Administration of Lansoprazole | 2: Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome is the Number of Days to Become Free of Narcotic Pain Medication.
Time Frame: 2 weeks
Population: as for baseline characteristics
Arm/Group | 1: Post-operative Administration of Lansoprazole | 2: Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: The Secondary Outcomes Are the Number of Days to be Free of Pain, the Number of Days to Return to Normal Activity Levels and the Number of Days to Return to Normal Fluid Intake.
Time Frame: 2 weeks
Population: as for baseline characteristics
Arm/Group | Lansoprazole | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The study was terminated due to low recruitment, since only one participant returned logbooks with data there are concerns with confidentiality therefore no data is being reported.
Description: The study was terminated due to low recruitment, since only one participant returned logbooks with data there are concerns with confidentiality therefore no data is being reported.
Arm/Group | 1: Post-operative Administration of Lansoprazole | 2: Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No